CLINICAL TRIAL: NCT01879592
Title: Molecular Phenotyping of Asthma in Sickle Cell Disease
Acronym: MoP-ASC
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Kathryn Blake, PharmD, Senior Research Scientist, Nemours Children's Clinic
Other Study IDs: 202349
Record Dates: First submitted 2013-04-12; First posted 2013-06-18 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Sickle Cell Disease; Asthma
Keywords: Sickle cell disease; Asthma; Metabolomics; Gene expression
MeSH Terms: conditions — Anemia, Sickle Cell; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood (RBC, WBC, DNA), urine, and saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Asthma + sickle cell disease: African American children affected with both sickle cell disease and asthma
- Sickle cell disease: African American children affected with sickle cell disease but who do not have asthma
- Asthma: African American children affected with asthma but without sickle cell disease
- Healthy control: African American children who are healthy with no chronic disease

SUMMARY:
Asthma and sickle cell disease each are serious medical problems. People with asthma have difficulty breathing, wheeze (a whistling noise when breathing), cough, produce sputum or phlegm, and have inflammation (swelling, irritation, redness) and narrowing of the bronchial tubes.

When a person has both asthma and sickle cell disease together, more serious medical problems can occur such as having acute chest syndrome and pain episodes more often. It is sometimes hard to diagnose asthma in a person with sickle cell disease because sickle cell disease can also cause lung problems.

The purpose of this study is to see if the investigators can better understand asthma when it occurs in a person who has sickle cell disease. The investigators will do this by taking a blood, urine, and saliva sample. The blood and urine samples will be analyzed for chemicals and DNA (genes). Certain genes can cause patients to have sickle cell disease or asthma. The investigators will use the saliva sample for future studies to compare the results from the blood testing with saliva. The investigator's long-term goal is to make sure people who have asthma and sickle cell disease are getting the best asthma treatments. The investigator's hypothesis is that the analysis of the blood, urine and saliva using a method called, metabolomics, may identify a unique asthma signature in children with sickle cell disease which may lead to targeted treatments.

DETAILED DESCRIPTION:
Asthma recently has been described as a disorder of multiple subphenotypes despite a common symptom presentation. These subphenotypes have differing molecular pathways and discovering these differences may lead to better diagnosis strategies and new treatments. Most studies investigating asthma pathways are driven by the scientist's own theories and experience and thus, are considered biased. Metabolomics, an exciting and innovative discipline, represents an unbiased, hypothesis free approach to defining a molecular phenotype of asthma.

Sickle cell disease is a common genetic disorder and there is ample evidence that asthma is a common co-morbidity with an asthma prevalence of 2% to 45% compared with 12.8% in African American children without sickle cell disease. Acute chest syndrome (ACS) contributes to the cause of death in up to 60% of deaths in sickle cell patients and there is a strong relationship between having asthma and the risk of developing ACS and an increased risk of death.

Metabolomics is the study of the entire repertoire of small molecules present in cells, tissues, organs and biological fluids that comprise the metabolome. Metabolomics measures the downstream products of protein, gene, and environmental interactions and importantly, comes closest to expressing phenotype, and provides the opportunity to explore gene by environment and gene by gene interactions. A systems biology approach using metabolomics has been advocated to better understand pulmonary disease.

Asthma in the sickle cell patient is likely to have a molecular fingerprint which can be distinguished from asthma in the non-sickle cell patient. The investigator's specific aim is to compare the urinary metabolomic profile of children with asthma and sickle cell disease to children without asthma who have sickle cell disease, and to a cohort of African American children with asthma but without sickle cell disease. The hypothesis is that children with asthma and sickle cell disease will have a unique metabolomic profile that will discriminate these patients from children with sickle cell disease who have respiratory dysfunction that is not asthma, and from children with asthma who do not have sickle cell disease.

The investigators will collect a single saliva, urine and blood specimen from children with asthma and sickle cell disease, children with sickle cell disease only, and African American children with asthma only for metabolomic analysis. A single urine sample will be collected from health African American children without any chronic diseases. Blood will be stored for a future study to compare metabolomic variability between blood and urine. The investigator's goal is to use this information to correctly identify children with asthma. These data will enhance the investigator's understanding of the mechanisms that underlie the molecular asthma phenotype in sickle cell disease, which should lead to more targeted treatment of asthma in sickle cell disease. The investigators long-term goal is to reduce the burden of asthma in the child with sickle cell disease (pain, ACS, and death) by using this innovative systems biology approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged 6 years old up to 21 years old
* Children with sickle cell disease with the genotype SS, SC, or S β 0 thal
* African American children with asthma who do not have sickle cell disease or sickle cell disease trait.
* African American children with no chronic disease
* Physician diagnosed asthma and atopy (of any asthma severity) plus a family history of asthma 89,90
* Patients whose controller respiratory medications and maintenance medications for sickle cell disease (e.g. hydroxyurea) have been unchanged for the previous 4 weeks

Exclusion Criteria:

* Patients who are current smokers
* Patients who had an inflammatory event related to sickle cell disease (pain episode, priapism, acute chest syndrome, urgent medical visit), asthma exacerbation, or respiratory infection within 1 month prior to the blood, saliva, and urine collection.
* Patients who are receiving chronic transfusion therapy and who have received a transfusion within 90 days prior to blood, saliva, and urine collection.
* Patients who have received treatment with a leukotriene synthesis inhibitor or a leukotriene modifier[montelukast (Singulair®)] within the 2 weeks prior to blood and urine collection.
* Women who are pregnant or lactating

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Three groups of 30 children each will be studied: Group 1, children with asthma and sickle cell disease; Group 2, children with sickle cell disease but without asthma; Group 3, control group of 30 African American children with asthma but without sickle cell disease ; Group 4, healthy control group of 25 African American children with no chronic disease. All children are seen at Nemours Children's Clinics in Jacksonville FL, Orlando FL, or Wilmington DE.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2011-06; Primary Completion 2016-02-28 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Metabolomic Principal Component Profile | Day 1
  Principal component analysis of differences in the variability in the metabolomic profile of children with asthma and sickle cell disease compared with children with sickle cell disease only and a cohort of African American children with asthma only and a cohort of African American children with no chronic disease.

SECONDARY OUTCOMES:
Placenta Growth Factor (PlGF) plasma concentrations | Day 1
  Differences in PlGF plasma concentrations in children with asthma and sickle cell disease compared with children with sickle cell disease only and a cohort of African American children with asthma only.
Messenger ribonucleic acid (mRNA) transcript levels | Day 1
  Differences in mRNA transcript levels of 5-lipoxygenase (ALOX5) and five-lipoxygenase activating protein (FLAP) genes in children with asthma and sickle cell disease compared with children with sickle cell disease only and a cohort of African American children with asthma only.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Blake, PharmD, Principal Investigator — Nemours Children's Clinic
Locations (3):
- United States (3):
  - Nemours Children's Clinic, Wilmington, Delaware
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Our consent documents did not include sharing of individual participant data